CLINICAL TRIAL: NCT01204346
Title: Mentalization - Based Treatment for Young People Presenting With Co-morbid Depression and Symptoms of Emerging Personality Disorder: Prospective Controlled Trial.
Brief Title: Mentalization - Based Treatment: Adolescents With Co-morbid Depression and Personality Disorder
Acronym: MBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North East London Foundation Trust (Other)
Responsible Party: Principal Investigator, Trudie Rossouw, Dr, North East London Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRossouw
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2011-07

CONDITIONS: Depression; Personality Disorder
Keywords: adolescents; MBT; depression; emerging personality disorder
MeSH Terms: conditions — Depression; Personality Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBT group (Experimental): mentalization based treatment program
  Interventions: Other: MBT
- Treatment as usual group (Active Comparator): treatment as usual group
  Interventions: Other: treatment as usual

INTERVENTIONS:
Other: MBT — The intervention consists of twice weekly individual MBT therapy, group therapy with an MBT focus and weekly MBFT, which is MBT for families. The treatment duration will be 6-8 weeks.
  Other Names: Psychotherapeutic program
  Arms: MBT group
Other: treatment as usual — less intensive and structured psychotherapeutic program
  Other Names: Psychotherapeutic program
  Arms: Treatment as usual group

SUMMARY:
Mentalisation based treatment (MBT) for young people with co-morbid depression and emerging personality disorder will be more effective in a day/inpatient setting than treatment as usual.

DETAILED DESCRIPTION:
Systematic literature review on outcomes with young people with depression and emerging personality disorder showed clear evidence that this group of young people are severely hampered and adult outcomes are strongly linked to both adult PD as well as adult psychiatric disturbance and lower levels of adult functioning. (Crawford et al, 2008; Kasen et al, 1999; Kasen et al, 2007; Lewinsohn et al, 1999) This argues very clearly for the need to diagnose young people presenting with co-morbid depression and emerging personality disorder in order to intervene and help these young people's struggles as it will prevent poor prognostic adult outcomes. There were no treatment programs that specifically focussed on the treatment of this co-morbid group in the literature. Several studies focussed on the treatment of depression alone and only one RCT focussed on the treatment of adolescent personality disorder (Chanen et al, 2007). In adult studies mentalization-based treatment programs were found to be effective ( as well as cost effective) in a day hospital setting for adults with personality disorder and depression (Bateman, et al, 2007) This study aims to conduct a control trial to test whether MBT will be more effective than TAU in this group. All cases will be tested on admission, at discharge and followed up at 2 years post discharge.

ELIGIBILITY:
Inclusion Criteria:

* all young people who are admitted to Brookside adolescent unit between the ages 12 - 17 presenting with depression and emerging personality disorder will be eligible

Exclusion Criteria:

* Young people with autistic spectrum disorders or severe learning disabilities.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2010-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Global assessment of functioning | 2 years post discharge
  Measures global functioning
Global assessment of functioning | within 1 week of admission
  measures level of functioning
global assessment of functioning | Average of 8 weeks
  measures level of functioning

SECONDARY OUTCOMES:
mood and feelings questionnaire | 2 years post discharge
  Assesses mood in terms of number of depressive symptoms
Mood and feelings questionnaire | Within 1 week of admission
  Assesses mood in terms of number of depressive symptoms
mood and feelings questionnaire | At average of 8 weeks
  Assesses mood in terms of number of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: trudie i rossouw, dr, Principal Investigator — North East London Foundation Trust
Locations (1):
- North East London Foundation Trust, Ilford, Essex, United Kingdom

REFERENCES:
- [Background] Bateman A, Fonagy P. Mentalization based treatment for borderline personality disorder. World Psychiatry. 2010 Feb;9(1):11-5. doi: 10.1002/j.2051-5545.2010.tb00255.x. PMID 20148147
- [Background] Bateman A, Fonagy P. Randomized controlled trial of outpatient mentalization-based treatment versus structured clinical management for borderline personality disorder. Am J Psychiatry. 2009 Dec;166(12):1355-64. doi: 10.1176/appi.ajp.2009.09040539. Epub 2009 Oct 15. PMID 19833787
- [Background] Crawford TN, Cohen P, First MB, Skodol AE, Johnson JG, Kasen S. Comorbid Axis I and Axis II disorders in early adolescence: outcomes 20 years later. Arch Gen Psychiatry. 2008 Jun;65(6):641-8. doi: 10.1001/archpsyc.65.6.641. PMID 18519822
- [Background] Kasen S, Cohen P, Skodol AE, Johnson JG, Brook JS. Influence of child and adolescent psychiatric disorders on young adult personality disorder. Am J Psychiatry. 1999 Oct;156(10):1529-35. doi: 10.1176/ajp.156.10.1529. PMID 10518162
- [Background] Kasen S, Cohen P, Skodol AE, First MB, Johnson JG, Brook JS, Oldham JM. Comorbid personality disorder and treatment use in a community sample of youths: a 20-year follow-up. Acta Psychiatr Scand. 2007 Jan;115(1):56-65. doi: 10.1111/j.1600-0447.2006.00842.x. PMID 17201867
- [Background] Lewinsohn PM, Rohde P, Klein DN, Seeley JR. Natural course of adolescent major depressive disorder: I. Continuity into young adulthood. J Am Acad Child Adolesc Psychiatry. 1999 Jan;38(1):56-63. doi: 10.1097/00004583-199901000-00020. PMID 9893417
- [Background] Chanen AM, McCutcheon LK, Jovev M, Jackson HJ, McGorry PD. Prevention and early intervention for borderline personality disorder. Med J Aust. 2007 Oct 1;187(S7):S18-21. doi: 10.5694/j.1326-5377.2007.tb01330.x. PMID 17908019
- See also: host NHS organisation — http://www.nelft.nhs.uk/